CLINICAL TRIAL: NCT04106388
Title: An Evaluation of Virtual Behavioral Health Integration Into Primary Care
Brief Title: Virtual Behavioral Health Integration
Acronym: VBHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00082499; 08-19-24E (Other: Atrium)
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2021-06

CONDITIONS: Depression; Substance Use Disorder; Anxiety
MeSH Terms: conditions — Depression; Substance-Related Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Locations offering the program are randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Behavioral Health Integration (Experimental): All patients who meet eligibility criteria at sites where the virtual behavioral health program is offered will be considered exposed to the intervention.
  Interventions: Behavioral: Virtual Behavioral Health Integration
- Usual Care - Behavioral Health (No Intervention): All patients who meet eligibility criteria at sites where the virtual behavioral health program is not offered will be considered exposed to usual care.

INTERVENTIONS:
Behavioral: Virtual Behavioral Health Integration — The virtual behavioral health integration program, implemented in primary care settings, is a structured mental illness treatment program that includes both behavioral treatment and counseling components aimed at reducing cost of care, developing and sustaining adaptive coping strategies, and improving short term acute care utilization.
  Arms: Virtual Behavioral Health Integration

SUMMARY:
The primary objective is to evaluate the effectiveness of the virtual behavioral health integration (VBHI) program compared to usual care, on reducing the total cost of care reimbursed from Medicare and value-based contracts within 90 days of a patient's primary care visit.

DETAILED DESCRIPTION:
To enhance the care of patients seen in the primary care setting, Atrium Health has designed a virtual behavioral health integration program. A behavioral health care team comprised of licensed clinicians (Behavioral Health Professionals), health coaches, a consulting psychiatric pharmacist and psychiatric providers follow patients for up to 3 months or more depending on patient need after their primary care office visit. This virtual behavioral health integration (VBHI) program is currently available in 36 Atrium Health primary care practices providing support to over 200 providers and medical residents. The Behavioral health Service line is expanding the program to additional primary care practices. Atrium Health and the Carolinas Physician Alliance is interested in evaluating the effectiveness of the program on reducing the total cost of care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Primary care office visit
* Have a Patient Health Questionnaire-9 (PHQ-9) and overall score >=10 or Question 9 >0
* Medicare or value-based contract associated with a patient in the past year at the time of the primary care visit.

Exclusion Criteria:

* A patient will contribute to the analysis once using their initial enrollment to either arm of the study.
* No insurance claim for the index primary care visit in the data warehouse upon evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5777 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Cost of Care | 90 days from a patient's primary care visit
  Total cost of care reimbursed from Medicare and value-based contracts

SECONDARY OUTCOMES:
Compare the 90-day acute care utilization rate after the index primary care visit | 90 days from a patient's primary care visit
  Does a patient have an inpatient, observation, or emergency department encounter after their primary care visit
Compare the 90-day primary care utilization rate after the index primary care visit | 90 days from a patient's primary care visit
  Does a patient have a primary care encounter after their primary care visit
pharmacy Cost of Care | 90 days from a patient's primary care visit
  Pharmacy related cost of care reimbursed from Medicare and value-based contracts

CONTACTS AND LOCATIONS:
Overall Officials: Jason Roberge, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (20):
- United States (20):
  - Albermarle Medical Services, Albemarle, North Carolina
  - Charlotte Medical Clinic Arboretum, Charlotte, North Carolina
  - North Charlotte Medical Specialists Huntersville, Charlotte, North Carolina
  - Mecklenburg Medical Group - Steele Creek, Charlotte, North Carolina
  - NorthEast Internal and Integrative Medicine, Concord, North Carolina
  - East Lincoln Primary Care, Denver, North Carolina
  - Riverwood Medical Associates, Gastonia, North Carolina
  - Ardsley Internal Medicine - Harrisburg, Harrisburg, North Carolina
  - Dove Internal Medicine Union West, Indian Trail, North Carolina
  - Indian Trail Family Medicine, Indian Trail, North Carolina
  - Kannapolis Internal Medicine, Kannapolis, North Carolina
  - Kings Mountain Internal Medicine, Kings Mountain, North Carolina
  - West Lincoln Family Medicine, Lincolnton, North Carolina
  - Dove Internal Medicine - Monroe, Monroe, North Carolina
  - Union Family Practice, Monroe, North Carolina
  - Mooresville Internal Medicine Associates, Mooresville, North Carolina
  - Oakboro Medical Services, Oakboro, North Carolina
  - Richfield Medical Services, Richfield, North Carolina
  - Shelby Family Practice, Shelby, North Carolina
  - Union Primary Care, Wesley Chapel, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT04106388/Prot_SAP_000.pdf